CLINICAL TRIAL: NCT05613491
Title: Intranasal Insulin Improves Postoperative Neurocognitive Disorders in Elderly Patients: a Multicenter, Randomized, Double-blind, Placebo-controlled Study
Brief Title: Intranasal Insulin Improves Postoperative Neurocognitive Disorders in Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Tang-Du Hospital (Other); Tongji Hospital (Other); Second Hospital of Shanxi Medical University (Other); LanZhou University (Other); Sichuan Provincial People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); 521 Hospital of NORINCO Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: XJTU1AF2022LSK-265
Record Dates: First submitted 2022-11-06; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Postoperative Neurocognitive Disorders
Keywords: postoperative neurocognitive disorders; Intranasal insulin
MeSH Terms: interventions — Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intranasal insulin group (Experimental): Before anesthesia induction, give the first insulin nasal spray, once per hour, 20 IU each time, until the end of the operation
  Interventions: Drug: Intranasal insulin
- Saline group (Placebo Comparator): Before anesthesia induction, give the equal volumes'saline nasal spray, once per hour, 20 IU each time, until the end of the operation
  Interventions: Drug: Intranasal saline

INTERVENTIONS:
Drug: Intranasal insulin — Put insulin injection into nasal special drug delivery device.Before anesthesia induction, give the first insulin nasal spray, once per hour, 20 IU each time, until the end of the operation
  Other Names: Insulin injection，H10890001,Jiangsu Wanbang Biochemical Medicine Group Co., Ltd
  Arms: Intranasal insulin group
Drug: Intranasal saline — Put 0.9% sodium chloride into nasal special drug delivery device.Before anesthesia induction, give the first equal volume saline nasal spray, once per hour, 20 IU each time, until the end of the operation
  Other Names: 0.9% sodium chloride，H20013250,Shanghai Baite Medical Supplies Co., Ltd
  Arms: Saline group

SUMMARY:
Postoperative neurocognitive disorders (PND) are common postoperative complication of central nervous system, leading to increased risk of the working ability loss after surgery, longer hospital stay, increased medical costs and increased surgical mortality. It is classified as perioperative neurocognitive disorders in mental disorders.Aging is an important demographic characteristic in China, and the elderly is also a population susceptible to PND. There is a lack of targeted prevention and control measures for PND. Central insulin resistance is an important mechanism of cognitive impairment in elderly patients, and exogenous supply of central insulin may be an important measure to improve PND. Compared with conventional subcutaneous and intravenous supply, intranasal insulin administration not only has little effect on blood glucose and insulin levels, but also enters the center through the blood-brain barrier easily and efficiently. Long-term use of intranasal insulin can improve the cognitive function of chronic diseases, but there is a lack of clinical studies on improving PND by intranasal insulin. This study will verify the effectiveness of intranasal insulin in the PND improvement of elderly patients.

DETAILED DESCRIPTION:
This study is intended to carry out a large sample, multicenter, double-blind, randomized, placebo, and controlled clinical study. Elderly non diabetes patients undergoing elective extrathoracic, breast, orthopedic, urinary, abdominal, and gynecological operations under general anesthesia are included. They are randomly divided into intranasal insulin group or saline group. Before anesthesia induction, they are given the first nasal spray, once per hour, 20 IU insulin or equal volume saline each time until the end of the operation. Follow up 1 day before operation, 1-7 days after operation, 30 days and 12 months respectively, and evaluate cognition with relevant scales. To verify that compared with the same volume of saline, intranasal insulin can reduce the incidence of postoperative delirium, the incidence of PND 1 year after surgery, and the related cognitive quantitative indicators of ApoE- ɛ4 Gene susceptibility, intraoperative EEG parameters, NfL, IL-6, IL-10, CRP and other biochemical indicators were used to explore the mechanism of intranasal insulin to improve PND.

ELIGIBILITY:
Inclusion Criteria:

* Patients under general anesthesia through oral intubation;
* Patients undergoing elective extrathoracic, breast, orthopaedic, urological, abdominal and gynecological operations;
* Age ≥ 65 years;
* Cardiac function grade I~II (NYHA standard), ASA grade I~III;
* Volunteer for anticipating study and sign an informed consent form;

Exclusion Criteria:

* Diabetes patients;
* Previous history of craniocerebral and spinal cord trauma, surgery, stroke, and inability to place electrodes on the head;
* History of nasal cavity stuffiness, epistaxis, rhinitis, and nasopharynx surgery; The operation position is prone and it is difficult to implement intranasal administration;
* Those who cannot cooperate with the assessment of the scale or have delirium before operation;
* Preoperative fasting blood glucose<4 mmol/L;
* Those who have participated in other clinical trials.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 438 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | 0-7 days after surgery
  Whether or not postoperative delirium happens

SECONDARY OUTCOMES:
Incidence of delayed neurocognitive recovery within 30 days after surgery | 0-30 days after surgery
  Whether or not delayed neurocognitive recovery happens
Incidence of neurocognitive disorders within 1 year after surgery | 30 day-1 year after surgery
  Whether or not neurocognitive disorders happens
The PND Incidence | 0 day-1 year after surgery
  Whether or not postoperative neurocognitive disorders happensevents after surgery
Intraoperative electroencephalogram parameters | Surgery day
  The intraoperative parameters recorded by electroencephalogram, including BIS occurrence time, the duration with PSI less than 25, spectrum analysis, power spectrum analysis.
the level of Neurocognitive biomarkers | 0 day-1 year after surgery
  Neurocognitive biomarkers includes amyloid-beta protein and tau protein.
ApoE-ε4 susceptibility | 1 day before surgery
  Whether or not carry ApoE-ε4

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Wang, MD,PHD, Study Chair — First Affiliated Hospital of Xian JiaotongUniversity
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: Yes
The research plan will not be made public until the research results are published
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Evered L, Silbert B, Knopman DS, Scott DA, DeKosky ST, Rasmussen LS, Oh ES, Crosby G, Berger M, Eckenhoff RG; Nomenclature Consensus Working Group. Recommendations for the nomenclature of cognitive change associated with anaesthesia and surgery-2018. Br J Anaesth. 2018 Nov;121(5):1005-1012. doi: 10.1016/j.bja.2017.11.087. Epub 2018 Jun 15. PMID 30336844
- [Background] Liu Y, Xiao W, Meng LZ, Wang TL. Geriatric Anesthesia-related Morbidity and Mortality in China: Current Status and Trend. Chin Med J (Engl). 2017 Nov 20;130(22):2738-2749. doi: 10.4103/0366-6999.218006. PMID 29133765
- [Background] Evered L, Scott DA, Silbert B, Maruff P. Postoperative cognitive dysfunction is independent of type of surgery and anesthetic. Anesth Analg. 2011 May;112(5):1179-85. doi: 10.1213/ANE.0b013e318215217e. Epub 2011 Apr 7. PMID 21474666
- [Background] Jayaraj RL, Azimullah S, Beiram R. Diabetes as a risk factor for Alzheimer's disease in the Middle East and its shared pathological mediators. Saudi J Biol Sci. 2020 Feb;27(2):736-750. doi: 10.1016/j.sjbs.2019.12.028. Epub 2019 Dec 26. PMID 32210695
- [Background] Li X, Run X, Wei Z, Zeng K, Liang Z, Huang F, Ke D, Wang Q, Wang JZ, Liu R, Zhang B, Wang X. Intranasal Insulin Prevents Anesthesia-induced Cognitive Impairments in Aged Mice. Curr Alzheimer Res. 2019;16(1):8-18. doi: 10.2174/1567205015666181031145045. PMID 30381076
- [Background] Chen Y, Dai CL, Wu Z, Iqbal K, Liu F, Zhang B, Gong CX. Intranasal Insulin Prevents Anesthesia-Induced Cognitive Impairment and Chronic Neurobehavioral Changes. Front Aging Neurosci. 2017 May 10;9:136. doi: 10.3389/fnagi.2017.00136. eCollection 2017. PMID 28539885
- [Background] Zhang Y, Dai CL, Chen Y, Iqbal K, Liu F, Gong CX. Intranasal Insulin Prevents Anesthesia-Induced Spatial Learning and Memory Deficit in Mice. Sci Rep. 2016 Feb 16;6:21186. doi: 10.1038/srep21186. PMID 26879001
- [Background] Claxton A, Baker LD, Hanson A, Trittschuh EH, Cholerton B, Morgan A, Callaghan M, Arbuckle M, Behl C, Craft S. Long-acting intranasal insulin detemir improves cognition for adults with mild cognitive impairment or early-stage Alzheimer's disease dementia. J Alzheimers Dis. 2015;44(3):897-906. doi: 10.3233/JAD-141791. PMID 25374101
- [Background] Benedict C, Hallschmid M, Schultes B, Born J, Kern W. Intranasal insulin to improve memory function in humans. Neuroendocrinology. 2007;86(2):136-42. doi: 10.1159/000106378. Epub 2007 Jul 20. PMID 17643054
- [Background] Chapman CD, Schioth HB, Grillo CA, Benedict C. Intranasal insulin in Alzheimer's disease: Food for thought. Neuropharmacology. 2018 Jul 1;136(Pt B):196-201. doi: 10.1016/j.neuropharm.2017.11.037. Epub 2017 Nov 24. PMID 29180222
- [Background] Benedict C, Hallschmid M, Hatke A, Schultes B, Fehm HL, Born J, Kern W. Intranasal insulin improves memory in humans. Psychoneuroendocrinology. 2004 Nov;29(10):1326-34. doi: 10.1016/j.psyneuen.2004.04.003. PMID 15288712
- [Background] Novak V, Milberg W, Hao Y, Munshi M, Novak P, Galica A, Manor B, Roberson P, Craft S, Abduljalil A. Enhancement of vasoreactivity and cognition by intranasal insulin in type 2 diabetes. Diabetes Care. 2014;37(3):751-9. doi: 10.2337/dc13-1672. Epub 2013 Oct 7. PMID 24101698
- [Background] Brunner YF, Kofoet A, Benedict C, Freiherr J. Central insulin administration improves odor-cued reactivation of spatial memory in young men. J Clin Endocrinol Metab. 2015 Jan;100(1):212-9. doi: 10.1210/jc.2014-3018. PMID 25337926